CLINICAL TRIAL: NCT01622504
Title: A Phase I Single Dose, Open Label, Randomized, Three Period Crossover Pilot Study to Compare the Pharmacokinetics, Safety and Tolerability of MVP005 Intranasal Spray With Intranasal Administration of Naloxone Solution for Injection in Healthy Adult Subjects
Brief Title: Naloxone Nasal Spray Pharmacokinetic Study
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mitovie Pharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MVP005-CLN-001
Record Dates: First submitted 2012-06-13; First posted 2012-06-19 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-06

CONDITIONS: Opioid Overdose
Keywords: Intranasal; nasal spray; opioid; overdose
MeSH Terms: conditions — Opiate Overdose; Drug Overdose | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Test Product Dose 1 (Experimental)
  Interventions: Drug: MVP005
- Test Product Dose 2 (Experimental)
  Interventions: Drug: MVP005
- Comparator Product (Active Comparator)
  Interventions: Drug: Naloxone hydrochloride solution for injection with mucosal atomization device

INTERVENTIONS:
Drug: MVP005 — 2 mg single dose administered intranasally
  Arms: Test Product Dose 1
Drug: MVP005 — 4 mg single dose administered intranasally
  Arms: Test Product Dose 2
Drug: Naloxone hydrochloride solution for injection with mucosal atomization device — 2 mg single dose administered intranasally
  Arms: Comparator Product

SUMMARY:
This study aims to compare the pharmacokinetics of naloxone when administered as the Mitovie nasal spray (Test Product) and as a solution for injection (Comparator Product) administered intranasally using a mucosal atomization device (MAD).

DETAILED DESCRIPTION:
Naloxone hydrochloride is currently only recommended and licensed for intravenous, intramuscular and subcutaneous administration. It has also been used by intranasal administration (off-label use) when the intravenous route is not suitable by administering the Solution for Injection using a mucosal atomization device (MAD). However, due to the volume of naloxone solution administered this way, some of it may be inadvertently swallowed and not absorbed into the nasal mucosa and the product requires administration by medically trained personnel. The study aims to investigate intranasal administration of naloxone using a more concentrated solution and a nasal delivery device.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* 18-60 50 years of age
* Provide written informed consent prior to completing any study specific procedure.
* Body Mass Index (BMI) range 18.5-30 kg/m2
* Clinically acceptable medical history, clinical laboratory evaluations, complete physical examination, vital signs and 12 lead ECG
* Using reliable contraception

Exclusion Criteria:

* Intranasal problems
* Taking prescribed or over the counter medications
* Intake of alcohol, methyl-xanthines or grapefruit or strenuous exercise concurrent with treatment.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Estimated)
Dates: Start 2012-06; Primary Completion 2012-07 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics | 0, 5, 10, 15, 20, 30 and 45 minutes and 1.00, 1.50, 2.00, 3.00, 4.00, 6.00, 8.00 and 12.00 hours for each arm
  Plasma concentration time profiles and area under the curve (AUC), maximum concentation (Cmax), Time to maximum concentration (Tmax), elimination rate constant (Kel) and terminal half life (t1/2)

SECONDARY OUTCOMES:
Number of subjects with adverse events | 14 days
  Continuous adverse event monitoring during the study with prompted assessments in the 12 hours post-dose
Physical Examination | 14 days
  Complete physical examination at screening and final follow-up and specific nasal examination post-dose
Vital signs | 14 days
  Vital signs at screening, final follow-up and pre- and post-dose
ECGs | 14 days
  ECGs at screening and final follow-up
Safety Laboratory Tests | 14 days
  Haematology, biochemistry and urinalysis at screening and final follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Abdullah Hiyari, MD, Principal Investigator — IPRC, Jordan
Locations (1):
- International Pharmaceutical Research Center (IPRC), Amman, Jordan